CLINICAL TRIAL: NCT06292104
Title: Multimodality Deep Phenotyping of Postural Orthostatic Tachycardia Syndrome (POTS), Aim 1
Brief Title: Phenotyping of Postural Orthostatic Tachycardia Syndrome (POTS)
Status: Recruiting | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Steven Vernino MD PhD, PROFESSOR, University of Texas Southwestern Medical Center
Other Study IDs: STU-2023-0589; 1R01HL166272-01A1 (NIH)
Record Dates: First submitted 2024-02-12; First posted 2024-03-04 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Postural Orthostatic Tachycardia Syndrome
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Serum, plasma and samples with DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- POTS (Postural Orthostatic Tachycardia Syndrome): Patients meeting clinical criteria for postural orthostatic tachycardia syndrome who meet other criteria for inclusion.
  Interventions: Diagnostic Test: multimodal diagnostic testing
- Healthy matched controls: Age and sex matched controls
  Interventions: Diagnostic Test: multimodal diagnostic testing

INTERVENTIONS:
Diagnostic Test: multimodal diagnostic testing — Serological testing, cardiac MRI, skin biopsy, cardiovascular testing, blood volume measurements

SUMMARY:
This is an observational study to deeply phenotype the disorder of POTS using multiple testing modalities.

DETAILED DESCRIPTION:
This comprehensive multimodality deep phenotyping will improve the diagnostic approach, inform the development of new treatments, and allow the targeting of therapies to specific POTS patients. The investigators will further identify the diagnostic tools, biomarkers, and clinical outcome measures most relevant to defining the disorder in clinical practice.

The specific aim is to (1) Define clinical POTS classifications from multimodal clinical and laboratory data, (2) address exercise tolerance in POTS using metabolomic assessments, (3) evaluate novel POTS-specific patient outcome measures and (4) evaluate one year outcome data for POTS

Specific research tests will include blood work (for immunophenotyping and neurohormonal assessments), autonomic function testing, skin biopsy (to evaluate intraepidermal nerve fiber density), CO (Carbon Monoxide) rebreathing (for quantitative measurement of plasma volume and red blood cell mass), patient surveys (to characterize symptom profile and disease impact). Blood biosamples will be stored as a repository for future research questions.

ELIGIBILITY:
Inclusion Criteria:

POTS Patients

* Age ≥ 14 years, able to provide informed consent (assent with parental consent for age < 18) and comply with procedures
* Meets consensus criteria for POTS: (1) sustained increase in heart rate ≥ 30 bpm above supine baseline within 10 min of quiet standing or upright tilt (≥ 40 bpm in individuals 12 to 19 years of age) OR sustained upright HR (heart rate) >120 bpm, (2) absence of orthostatic hypotension, (3) symptoms with standing that improve with sitting or lying down, (4) resting supine heart rate < 100 bpm, (5) orthostatic symptoms present for at least 6 months
* Stable oral medication regimen for at least 14 days

Non-POTS Control Patients

* Healthy women, age 18 - 30 years, able to provide informed consent and comply with study procedures
* Does NOT meet consensus criteria for postural tachycardia syndrome
* No symptoms of orthostatic intolerance or dysautonomia. No history of other major medical disorder
* Resting supine heart rate < 100 bpm

Exclusion Criteria:

None of the following exclusion criteria:

* Use of amphetamine-type stimulants, diuretics, selective norepinephrine reuptake inhibitor, anticholinergic medications (including tricyclic antidepressant medications), fludrocortisone, desmopressin in past 14 days
* Use of other autonomic drugs (adrenergic agents, pyridostigmine, droxidopa, triptans, ivabradine) in past 48 hours
* Currently receiving IVIG (Intravenous immunoglobulin), subcutaneous IgG (Immunoglobulin G), or any investigational medication (in past year)
* Infusion of iv fluids in past 7 days
* History or evidence of another condition explaining symptoms or orthostatic tachycardia (e.g. structural heart disease, CSF (Cerebrospinal fluid) hypovolemia, or severe traumatic brain injury)

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: POTS patients and Normal Control
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2024-03-05 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Phenotyping POTS | 2 weeks
  Assignment of participant to a phenotypic group(s) based on analysis of multimodal data
Natural history | 1 year
  Patient reported functional and subjective change. Surveys including COMPASS31 (Composite Autonomic Symptom Score-31) on a score of 0-100. Higher scores indicate more severe autonomic symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Steven Vernino, MD PhD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Raj SR, Bourne KM, Stiles LE, Miglis MG, Cortez MM, Miller AJ, Freeman R, Biaggioni I, Rowe PC, Sheldon RS, Shibao CA, Diedrich A, Systrom DM, Cook GA, Doherty TA, Abdallah HI, Grubb BP, Fedorowski A, Stewart JM, Arnold AC, Pace LA, Axelsson J, Boris JR, Moak JP, Goodman BP, Chemali KR, Chung TH, Goldstein DS, Darbari A, Vernino S. Postural orthostatic tachycardia syndrome (POTS): Priorities for POTS care and research from a 2019 National Institutes of Health Expert Consensus Meeting - Part 2. Auton Neurosci. 2021 Nov;235:102836. doi: 10.1016/j.autneu.2021.102836. Epub 2021 Jun 30. PMID 34246578
- [Background] Bryarly M, Phillips LT, Fu Q, Vernino S, Levine BD. Postural Orthostatic Tachycardia Syndrome: JACC Focus Seminar. J Am Coll Cardiol. 2019 Mar 19;73(10):1207-1228. doi: 10.1016/j.jacc.2018.11.059. PMID 30871704